CLINICAL TRIAL: NCT02252471
Title: Choices-Teen: A Bundled Risk Reduction Intervention for Juvenile Justice Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Danielle Parrish, Assistant Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1R03DA034099-01 (NIH)
Record Dates: First submitted 2014-09-20; First posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Alcohol Use; Smoking; Contraception; HIV
Keywords: alcohol-exposed pregnancy; nicotine-exposed pregnancy; tobacco-exposed pregnancy; alcohol; contraception; smoking; pregnancy; HIV; prevention
MeSH Terms: conditions — Alcohol Drinking; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Choices-Teen Intervention (Experimental): A three session intervention with two counseling sessions with a master's level therapist and a counseling session with a physician. The counseling with the master's level therapist utilizes a motivational interviewing approach to encourage changes in alcohol use, contraceptive use, smoking and HIV risk behaviors. This part of the intervention (a) provides norms-based-but personalized-feedback; (b) encourages participating in the smoking cessation program; (c) increases motivation to change each of the target behaviors; (d) decreases temptation to engage in risk behaviors; (e) increases confidence to avoid risk behaviors; and (f) develops a personalized, tailored change plan. The physician session provides individualized contraception and HIV risk reduction counseling.
  Interventions: Behavioral: Choices-Teen

INTERVENTIONS:
Behavioral: Choices-Teen — Choices-Teen participants in this condition will receive two brief motivational-interviewing-based counseling sessions, and one counseling session with a physician.

SUMMARY:
This pilot study will: 1) demonstrate the feasibility of delivering CHOICES-TEEN with master's level mental health professionals within a juvenile justice setting; 2) determine acceptance of CHOICES-TEEN as measured by client adherence, retention, and treatment satisfaction; and 3) assess client improvement at 3-month follow-up (e.g., reduction of risk of HIV, nicotine-exposed pregnancy, and alcohol-exposed pregnancy).

DETAILED DESCRIPTION:
The overall objective of this study is to assess the feasibility and promise of an adapted CHOICES preconception intervention (CHOICES-TEEN) in reducing the risk of HIV, nicotine-exposed pregnancy (NEP), and alcohol-exposed pregnancy (AEP) in adolescent females on intensive community probation. The current study posits that a two-session CHOICES intervention adapted to target multiple bundled health risks-AEP, NEP, and HIV-will be feasible, acceptable, and promising in reducing these risks among females on community-based juvenile probation. This study will: Aim 1: Modify the efficacious CHOICES preconception intervention to target the prevention of HIV, AEP, and NEP. The result will be a two session individual intervention (CHOICES-TEEN) and accompanying therapy manual based on the Transtheoretical Model (TTM) and Motivational Interviewing. Aim 2: Conduct a one-arm feasibility trial with females in the juvenile justice system to assess the promise of CHOICES-TEEN. This pilot study will: 1) demonstrate the feasibility of delivering CHOICES-TEEN with master's level mental health professionals within a juvenile justice setting; 2) determine acceptance of CHOICES-TEEN as measured by client adherence, retention, and treatment satisfaction; and 3) assess client improvement at 3-month follow-up (e.g., reduction of risk of HIV, NEP, and AEP). This study will inform subsequent Stage II/III behavioral intervention studies and contribute to a missing, fundamental element in the knowledge base - further understanding of the feasibility of targeting bundled health risks in high-risk adolescents, and the potential promise of a gender-specific intervention for this population.

ELIGIBILITY:
Inclusion Criteria:

* Have had vaginal intercourse with a male in the last 90 days
* Inconsistent/ineffective contraception use
* Inconsistent/ineffective condom use
* Drinking at risk levels
* Smoking
* Available for the follow-up period

Exclusion Criteria:

* Pregnant
* Infertile
* Insufficient locator information
* Language other than English

Ages: 14 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2012-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Risk of alcohol-exposed pregnancy | 3 months
  Timeline Followback Interview
Risk of nicotine-exposed pregnancy | 3 months
  Timeline Followback Interview
HIV risk | 3 months
  Timeline Followback Interview

SECONDARY OUTCOMES:
Excessive alcohol consumption | 3 months
  AUDIT Scale
Psychological distress and symptoms | 3 months
  Brief Symptom Inventory -18
Pros and cons of engaging in health risk behaviors (alcohol, smoking, HIV) | 3 months
  Decisional Balance Scale
Experiential and behavioral processes of change for health risk behaviors (alcohol, smoking, HIV) | 3 months
  Processes of Change Questionnaire
Temptation to engage in health risk behaviors (alcohol, smoking, HIV) | 3 months
  Temptation Scale
Confidence/self-efficacy to not engage in health risk behaviors (alcohol, smoking, HIV) | 3 months
  Confidence Scale

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E Parrish, Ph.D., Principal Investigator — University of Houston